CLINICAL TRIAL: NCT04622163
Title: Department of Medicine Secondary Mentoring Program Evaluation
Brief Title: Secondary Mentoring Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P001561
Record Dates: First submitted 2020-10-04; First posted 2020-11-09 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secondary Mentor Plus Career Development Resources (Experimental): Subjects will be assigned a secondary mentor for 6 months. Subjects will also receive career development resources.
  Interventions: Other: Secondary Mentor; Other: Career Development Resources
- Career Development Resources Alone (Other): Subjects will not be assigned a secondary mentor. Subjects will receive career development resources only.
  Interventions: Other: Career Development Resources

INTERVENTIONS:
Other: Secondary Mentor — Subjects will be matched with a secondary mentor from the Department of Medicine for 6 months. Mentors and mentees are expected to hold one-on-one meetings monthly for the first 3 months followed by at least once every 3 months thereafter.
  Arms: Secondary Mentor Plus Career Development Resources
Other: Career Development Resources — Subjects will receive career development resources.

SUMMARY:
Mentorship is essential to job satisfaction and promotion among academic physicians, and literature suggests that a single mentor is rarely sufficient. The investigators are studying whether implementation of a secondary mentorship program among physicians at their institution leads to improved job satisfaction over 6 months.

ELIGIBILITY:
Inclusion Criteria:

Physician employed as full-time faculty in the Massachusetts General Hospital Department of Medicine.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Job satisfaction | 6 months
  Job satisfaction is measured by the following question on a questionnaire developed by the investigators: "Overall how satisfied are you with your current position?" Responses are on a 5-point Likert scale (very unsatisfied, unsatisfied, neither, satisfied, very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States